CLINICAL TRIAL: NCT02791529
Title: Scalpel Versus Electrocautery for Surgical Skin Incision in Open Carpal Tunnel Release - Randomized, Controlled Open-Label Trial
Brief Title: Scalpel Versus Electrocautery for Surgical Skin Incision in Open Carpal Tunnel Release
Acronym: OCTR-Electro
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Intervention was inferior in pilot trial.
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYKS/OCTR-Electro/1-2
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Electrocoagulation; Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scalpel (Active Comparator): Skin incision performed by scalpel
  Interventions: Procedure: Scalpel
- Electrocautery (Experimental): Skin incision performed by electrocautery
  Interventions: Procedure: Electrocautery

INTERVENTIONS:
Procedure: Electrocautery — Skin incision performed by electrocautery
  Arms: Electrocautery
Procedure: Scalpel — Skin incision performed by scalpel
  Arms: Scalpel

SUMMARY:
The use of electrocautery for surgical skin incision in general surgery is known to decrease post-operative pain. This study compares the use of scalpel and electrocautery for surgical skin incision in open carpal tunnel release (OCTR).

DETAILED DESCRIPTION:
The use of electrocautery for surgical skin incision in general surgery is known to decrease post-operative pain. This study compares the use of scalpel and electrocautery for surgical skin incision in open carpal tunnel release (OCTR).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years
* Scheduled to undergo open carpal tunnel release (OCTR) by a study group member
* Gives informed consent
* diagnosis of chronic carpal tunnel syndrome

Exclusion Criteria:

* -Any current underlying systemic illness or condition that may affect wound healing (e.g. diabetes or chronic vascular disease)
* History of severe systemic or focal illness (e.g. previous myocardial infarction, chronic obstructive pulmonary disease)
* Chronic skin condition in the affected upper limb (e.g. psoriasis)
* Pregnancy
* Inability to comprehend the consent form (in Finnish) or inability to give consent
* Previous surgery or scar in the palmar aspect of the affected wrist
* Recurrent carpal tunnel syndrome
* Previous significant trauma of the affected upper extremity (including distal radius fracture) or suspicion of acute onset carpal tunnel syndrome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Pain on visual analogue scale | First postoperative day

IPD SHARING:
Plan to Share IPD: No